CLINICAL TRIAL: NCT00332046
Title: A Double-Blind, Randomized, Placebo-Controlled, Double-Dummy, Parallel Group, fMRI Study Comparing BOLD Activation Patterns Before and After 12 Weeks of Treatment With Placebo, Comparator and GW679769 in Subjects With Social Anxiety Disorder (SAD).
Brief Title: fMRI Study Comparing BOLD Activation Patterns Using GW679769 In Subjects With Social Anxiety Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NKF10015
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Social Anxiety Disorder
Keywords: fMRI placebo GW679769 Social Anxiety Disorder SAD
MeSH Terms: conditions — Phobia, Social | interventions — casopitant

INTERVENTIONS:
Drug: GW679769

SUMMARY:
Evidence suggests the use of neuroimaging to detect therapeutic effects of anxiolytic treatment when appropriate cognitive-emotional tasks are use to activate the emotional brain neurocircuitry believed to be involved in the core symptoms of the disease.

ELIGIBILITY:
Inclusion criteria:

* Primary diagnosis of Social Anxiety Disorder.
* Willing to restrict alcohol to a limited intake.

Exclusion criteria:

* History of schizophrenia, schizoaffective disorder or a bipolar disorder.
* Left-handed.
* Suffer from claustrophobia.
* Any reason why subject could not go into the fMRI, for example have metal implants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57
Dates: Start 2006-01

PRIMARY OUTCOMES:
Change in images of the brain, when stimulated, after once daily dosing for 12 weeks with GW679769, comparator or placebo in subjects with SAD.

SECONDARY OUTCOMES:
Blood levels of GW679769 and comparator at the Week 1 and Week 12 Change in clinical rating scales from baseline to Week 12 Safety & tolerability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, La Jolla, California, United States